CLINICAL TRIAL: NCT05837572
Title: Development of the Leeds Food Preference Questionnaire in Spanish: Sensitivity and Reproducibility of Liking and Wanting for Food in Fasted and Fed States
Brief Title: Development of the Leeds Food Preference Questionnaire in Spanish
Acronym: ES-LFPQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Principal Investigator, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ES-LFPQ Project
Record Dates: First submitted 2023-03-28; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Fasting; Fed
MeSH Terms: conditions — Fasting; Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Intervention Model Description: Participants are involved in two identical trials where they complete the ES-LFPQ under fasted and fed states (immediately after a standardised meal), at least one week apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Other): Each participant will attend the laboratory twice to perform two identical trials in order to asses validity (first trial) and reproducibility (second trial)
  Interventions: Other: Standardized meal

INTERVENTIONS:
Other: Standardized meal — Assessment of the validity of the ES-LFPQ: Each participant will complete the ES-LFPQ in before (fasted state) and after a standardized meal (fed state).
  Evaluation of the reproducibility of the ES-LFPQ: With at least one week of difference between tests, each participant will repeat the same protocol performed in the previous visit and under the same conditions.

SUMMARY:
The Leeds Food Preference Questionnaire (LFPQ) is a computer-based task used to measure reward responses and preferences for images of food. The present study aims to develop a Spanish version of the LFPQ (ES-LFPQ) by examining its validity and repeatability under fasted and fed states.

DETAILED DESCRIPTION:
The Leeds Food Preference Questionnaire (LFPQ) is a computer-based task for measuring reward responses (liking/wanting) and preferences for images of food. There are no cultural adaptation studies for the Spanish population to date in order to address its validity and repeatability in a test-retest design. The present study aim to develop a Spanish version of the LFPQ (ES-LFPQ), examine its outcomes under fasted and fed states; and test its reproducibility after one week.

An online survey containing foods that were either low-fat sweet, high-fat sweet, low-fat savoury or high-fat savoury was first conducted among a sample of 96 Spanish adults (60.4 % women) to develop and validate a culturally appropriate food image database. 50 participants (25 men and 25 women) will participate in two identical trials where they will completed the ES-LFPQ under fasted and fed states (immediately after a standardised meal), at least one week apart.

ELIGIBILITY:
Inclusion Criteria:

* Being able to understand instructions, programs and questionnaires.
* Being able to recognize the foods presented in at least 4 of the 5 photographs available for each category that make up the ES-LFPQ.
* Living in Spain for at least 2 years

Exclusion Criteria:

* Being intolerant, allergic and/or having an aversion to the foods contained in the standardized meal.
* Never eat the foods presented in at least 4 of the 5 photographs available for each category that make up the ES-LFPQ

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Explicit liking | 60 minutes
  The sensory pleasure elicited by contact with food. Measured with 0 to 100-mm visual analogue scale in response to the question "How pleasant would it be to taste some of this food now?" where 0 means "Not at all" and 100 means "Extremely"
Explicit wanting | 60 minutes
  The motivation to consume a specific food manifesting explicitly (conscious and subjective). Measured with 0 to 100-mm visual analogue scale in response to the question "How much do you want some of this food now?" where 0 means "Not at all" and 100 means "Extremely"
Implicit wanting | 60 minutes
  The motivation to consume a specific food manifesting implicitly (unconscious). Measured by punctuation on questionnaire ES-LFPQ. The score assigned to a specific food category based on a forced choice between pairs of food options and taking into account reaction time, in response to the question "Which food do you desire to consume the most at present?". A positive score indicates a greater preference for a given food category relative to the alternatives in the task and a negative score indicates the opposite. A score of zero would indicate that the category is equally preferred.
Relative preference | 60 minutes
  The preference of a food in comparison with another food. Measured by punctuation on questionnaire ES-LFPQ. The score assigned to a specific food category based on a forced choice between pairs of food options in response to the question "Which food do you desire to consume the most at present?". A positive score indicates a greater preference for a given food category relative to the alternatives in the task and a negative score indicates the opposite. A score of zero would indicate that the category is equally preferred.
Fat appeal bias | 60 minutes
  Bias scores for food fat content (high or low) computed by subtracting the mean low-fat scores from the mean high-fat scores. Positive values indicate a preference for high-fat, negative values indicate a preference for low fat and a score of 0 indicates an equal preference between fat content.
Taste appeal bias | 60 minutes
  Bias scores for food taste (savoury or sweet) computed by subtracting the mean savoury scores from the mean sweet scores. Positive values indicate a preference for sweet foods, negative values indicate a preference for savoury foods and a score of 0 indicates an equal preference between taste categories

SECONDARY OUTCOMES:
Hunger | 60 minutes
  The subjective sensation described as the primary motivation to eat. Measured with 0 to 100-mm visual analogue scale in response to the question "How hungry do you feel now?" where 0 means "Not at all" and 100 means "Extremely"
Fullness | 60 minutes
  The degree of satisfaction and/or fullness following food consumption. Measured with 0 to 100-mm visual analogue scale in response to the question "How full do you feel now?" where 0 means "Not at all" and 100 means "Extremely"

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada - Instituto Mixto Universitario Deporte y Salud, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided